CLINICAL TRIAL: NCT03586687
Title: Clinical Outcomes Following Randomization of Steroid Concentration in Patients With Glenohumeral Osteoarthritis
Brief Title: Osteoarthritis Shoulder Injection Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient rate of accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Cayce Onks, Assistant Professor of Family and Community Medicine and Orthopedics and Rehabilitation, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00008490
Record Dates: First submitted 2018-06-21; First posted 2018-07-13 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: Ultrasound guided injection
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 20 mg Triamcinolone with 3cc of 1% Lidocaine (Active Comparator): 20mg Triamcinolone with 3cc of 1% Lidocaine
  Interventions: Drug: Triamcinolone
- 40 mg Triamcinolone with 3cc of 1% Lidocaine (Active Comparator): 40mg Triamcinolone with 3cc of 1% Lidocaine
  Interventions: Drug: Triamcinolone
- 80 mg Triamcinolone with 3cc of 1% Lidocaine (Active Comparator): 80mg Triamcinolone with 3cc of 1% Lidocaine
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — Ultrasound guided glenohumeral shoulder joint injection

SUMMARY:
The purpose of this study is to determine the most effective intraarticular steroid dose for the treatment of glenohumeral osteoarthritis. The investigators aim to randomize patients into low, medium, and high dose groups of injectable corticosteroids as these doses are typically used in the standard of care for our patients. To date there has been no study to evaluate which dose is most efficient with the fewest side effects for glenohumeral osteoarthritis. The investigators objective will be to provide ultrasound guided intraarticular glenohumeral injections of these randomized concentrations and to evaluate pain and function before and following injection with the Shoulder Pain and Disability Index (SPADI). The investigators hypothesize that the low dose steroid will provide equivalent improvement of the pain and function to the medium and high doses, while minimizing side effects.

DETAILED DESCRIPTION:
Osteoarthritis (OA) affects 54.4 million US adults and 23.7 million (43.5%) have arthritis-attributable activity limitation. As the condition progresses, pain and functional disability increase. Patients usually begin treatment with conservative measures including physical therapy and administration of nonsteroidal anti-inflammatory drugs before obtaining a corticosteroid injection. Corticosteroid injections have a patient-specific duration that often provide relief for a month before the effects begin to taper with most individuals returning to baseline by 2-3 months post injection.

Unfortunately, data on intraarticular injections is not robust and primarily focused on hip, knee, and disease processes rather than the glenohumeral joint. For example, steroid concentrations have been studied in adhesive capsulitis, where 20 and 40mg of triamcinolone acenotide were used with no statistical significance between the two. When a placebo was added, both doses were better than the placebo, but once again no difference was seen between the two steroid concentrations. Another study, looking at knee osteoarthritis, found that high dose steroids had a larger effect on duration, but other studies have shown no difference in duration between the 40mg and 80mg concentration of triamcinolone acetonide.

Intraarticular injections do have adverse effects. Similar to steroids taken orally or intravenously, intraarticular injections have a similar side effect profile. Fortunately, intraarticular injections are localized, by the nature of the procedure, and the chances of experiencing a significant side effect is rare. The most common side effects are steroid flare, allergic reaction, facial erythema, hypo-pigmentation, fat pad necrosis, cutaneous atrophy, and a transient increase in blood glucose. Some of the rare side effects have been seen in case reports include idiopathic central serous chorioretinopathy, decrease in breast milk production, sepsis, tendon rupture, and cataracts. In addition, the administration of steroid injections are limited to being done every three months due to risk of weakening tendons, and acceleration of cartilage loss.

There is a void of literature for understating the ideal injectable steroid concentrations in glenohumeral osteoarthritis. Because of this, providers who perform intraarticular injections tend to perform them based on prior training experience or anecdotal evidence. We aim to evaluate the ideal steroid concentration that will maximize treatment effect for glenohumeral osteoarthritis, but at the same time minimize side effects, and better train our future providers.

ELIGIBILITY:
Inclusion Criteria:

* An X-ray within a year with Radiographic evidence of OA
* 18 years of age or older
* Clinical diagnosis established due to symptoms that will include pain attributed to glenohumeral osteoarthritis, pain with range of motion, and/or functional limitations longer than 3 months.

Exclusion Criteria:

* Previous guided steroid injection of the glenohumeral joint within 3 months
* Previous diagnosis of inflammatory arthritis, rotator cuff tear, or immunocompromised
* Previous shoulder surgery
* Allergy to steroid or lidocaine
* A Kellgren and Lawrence classification of 1 or less on radiograph
* Non-English Speaking
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cayce Onks, DO, Principal Investigator — Penn State Hershey Medical Cen
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour KE, Helmick CG, Boring M, Brady TJ. Vital Signs: Prevalence of Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation - United States, 2013-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 10;66(9):246-253. doi: 10.15585/mmwr.mm6609e1. PMID 28278145
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Godwin M, Dawes M. Intra-articular steroid injections for painful knees. Systematic review with meta-analysis. Can Fam Physician. 2004 Feb;50:241-8. PMID 15000335
- [Background] Arroll B, Goodyear-Smith F. Corticosteroid injections for osteoarthritis of the knee: meta-analysis. BMJ. 2004 Apr 10;328(7444):869. doi: 10.1136/bmj.38039.573970.7C. Epub 2004 Mar 23. PMID 15039276
- [Background] Gaujoux-Viala C, Dougados M, Gossec L. Efficacy and safety of steroid injections for shoulder and elbow tendonitis: a meta-analysis of randomised controlled trials. Ann Rheum Dis. 2009 Dec;68(12):1843-9. doi: 10.1136/ard.2008.099572. Epub 2008 Dec 3. PMID 19054817
- [Background] Kim YS, Lee HJ, Lee DH, Choi KY. Comparison of high- and low-dose intra-articular triamcinolone acetonide injection for treatment of primary shoulder stiffness: a prospective randomized trial. J Shoulder Elbow Surg. 2017 Feb;26(2):209-215. doi: 10.1016/j.jse.2016.09.034. Epub 2016 Nov 30. PMID 27914846
- [Background] Yoon SH, Lee HY, Lee HJ, Kwack KS. Optimal dose of intra-articular corticosteroids for adhesive capsulitis: a randomized, triple-blind, placebo-controlled trial. Am J Sports Med. 2013 May;41(5):1133-9. doi: 10.1177/0363546513480475. Epub 2013 Mar 18. PMID 23507791
- [Background] Popma JW, Snel FW, Haagsma CJ, Brummelhuis-Visser P, Oldenhof HG, van der Palen J, van de Laar MA. Comparison of 2 Dosages of Intraarticular Triamcinolone for the Treatment of Knee Arthritis: Results of a 12-week Randomized Controlled Clinical Trial. J Rheumatol. 2015 Oct;42(10):1865-8. doi: 10.3899/jrheum.141630. Epub 2015 Aug 1. PMID 26233499
- [Background] Intra-articular injections for osteoarthritis of the knee. Med Lett Drugs Ther. 2006 Mar 27;48(1231):25-7. No abstract available. PMID 16554699
- [Background] Smuin DM, Seidenberg PH, Sirlin EA, Phillips SF, Silvis ML. Rare Adverse Events Associated with Corticosteroid Injections: A Case Series and Literature Review. Curr Sports Med Rep. 2016 May-Jun;15(3):171-6. doi: 10.1249/JSR.0000000000000259. No abstract available. PMID 27172081
- [Background] McAlindon TE, LaValley MP, Harvey WF, Price LL, Driban JB, Zhang M, Ward RJ. Effect of Intra-articular Triamcinolone vs Saline on Knee Cartilage Volume and Pain in Patients With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1967-1975. doi: 10.1001/jama.2017.5283. PMID 28510679
- [Background] Kegel G, Marshall A, Barron OA, Catalano LW, Glickel SZ, Kuhn M. Steroid injections in the upper extremity: experienced clinical opinion versus evidence-based practices. Orthopedics. 2013 Sep;36(9):e1141-8. doi: 10.3928/01477447-20130821-15. PMID 24025004
- [Derived] Onks C, Weaver L, Latorre J, Silvis M, Berg A, Phillips S, Loeffert J, French C, Armstrong A. The most effective corticosteroid dose in the treatment of glenohumeral osteoarthritis: Feasibility pilot and protocol for double blinded randomized controlled trial. Osteoarthr Cartil Open. 2024 May 9;6(3):100484. doi: 10.1016/j.ocarto.2024.100484. eCollection 2024 Sep. PMID 38800822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mg Triamcinolone With 3cc of 1% Lidocaine | 40 mg Triamcinolone With 3cc of 1% Lidocaine | 80 mg Triamcinolone With 3cc of 1% Lidocaine
Started | 6 | 9 | 4
Completed | 6 | 9 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 20 mg: 20mg Triamcinolone with 3cc of 1% Lidocaine
  Triamcinolone: Ultrasound guided glenohumeral shoulder joint injection
- 40 mg: 40mg Triamcinolone with 3cc of 1% Lidocaine
  Triamcinolone: Ultrasound guided glenohumeral shoulder joint injection
- 80 mg: 80mg Triamcinolone with 3cc of 1% Lidocaine
  Triamcinolone: Ultrasound guided glenohumeral shoulder joint injection
- Total: Total of all reporting groups
Arm/Group | 20 mg | 40 mg | 80 mg | Total
Number analyzed (Participants) | 6 | 9 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.67 (12.26) | 69.33 (6.93) | 64.50 (12.29) | 66.53 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 4 | 5 | 1 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall SPADI Scores at Baseline Compared to 2,4, and 6 Months.
Description: The Shoulder Pain and Disability Index (SPADI) measures current shoulder pain and disability using a 13 item assessment. Scores range from 0-100 with higher scores indicating greater impairment or disability
Time Frame: baseline, 2, 4, and 6 months. Baseline SPADI score was collected prior to injection.
Population: Difference in subjects analyzed for all arms was due to the need of subsequent treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20 mg Triamcinolone With 3cc of 1% Lidocaine | 40 mg Triamcinolone With 3cc of 1% Lidocaine | 80 mg Triamcinolone With 3cc of 1% Lidocaine
Number analyzed (Participants) | 6 | 9 | 4
score on a scale
  Baseline SPADI Score | 58.17 (17.88) | 60.67 (17.91) | 44.50 (18.34)
  2 month SPADI Score: number analyzed (Participants) | 5 | 9 | 4
  2 month SPADI Score | 30.60 (22.60) | 48.67 (22.01) | 22.25 (19.97)
  4 month SPADI Score: number analyzed (Participants) | 5 | 8 | 3
  4 month SPADI Score | 44.80 (30.11) | 51.12 (27.53) | 35.67 (34.43)
  6 month SPADI Score: number analyzed (Participants) | 5 | 7 | 2
  6 month SPADI Score | 44.60 (25.60) | 57.71 (18.62) | 26.00 (7.07)

2. Primary Outcome: Assess Reactions to the Steroid
Description: Adverse events will only include those that are determined to be related to steroid Adverse Reactions to the Steroid are reported as combined for all the participants and not at the per-participant level.
Time Frame: baseline, 2, 4, and 6 months. Baseline data was collected at 2wks post injection phone call.
Measure: Number; unit: Reactions
Arm/Group | 20 mg Triamcinolone With 3cc of 1% Lidocaine | 40 mg Triamcinolone With 3cc of 1% Lidocaine | 80 mg Triamcinolone With 3cc of 1% Lidocaine
Number analyzed (Participants) | 6 | 9 | 4
Reactions
  Baseline | 1 | 2 | 0
  2 month follow up | 0 | 0 | 0
  4 month follow up | 0 | 0 | 0
  6 month follow up | 0 | 0 | 0

3. Secondary Outcome: Rate of Shoulder Arthroplasty Following Injection
Description: Shoulder arthroplasty is defined as total shoulder replacement
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg Triamcinolone With 3cc of 1% Lidocaine | 40 mg Triamcinolone With 3cc of 1% Lidocaine | 80 mg Triamcinolone With 3cc of 1% Lidocaine
Number analyzed (Participants) | 6 | 9 | 4
Participants | 3 | 1 | 1

4. Secondary Outcome: Change in Overall SPADI Scores for Those Receiving Shoulder Arthroplasty at 1 Year
Description: as for outcome 1
Time Frame: 12 months
Population: Subjects who underwent shoulder arthroplasty by/at 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20 mg Triamcinolone With 3cc of 1% Lidocaine | 40 mg Triamcinolone With 3cc of 1% Lidocaine | 80 mg Triamcinolone With 3cc of 1% Lidocaine
Number analyzed (Participants) | 1 | 1 | 1
score on a scale | 2 (NA) — Standard Deviation is not calculable for 1 participant | 12 (NA) — Standard Deviation is not calculable for 1 participant | 4 (NA) — Standard Deviation is not calculable for 1 participant

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months
Arm/Group | 20 mg | 40 mg | 80 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 2/9 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg (N=6) | 40 mg (N=9) | 80 mg (N=4)
Steroid flare (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial flushing (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Target enrollment was not reached due to the COVID pandemic. The secondary outcome measure involving SPADI at 12 months were not collected due to COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT03586687/Prot_SAP_000.pdf